CLINICAL TRIAL: NCT01840150
Title: A Single-center Study to Evaluate the Feasibility of a Novel NA-NOSE for Monitoring Response to and Detecting Recurrence After Surgery or Radiation in Early Stage Lung Cancer
Brief Title: Study to Evaluate NA-NOSE for Monitoring and Detecting Recurrence in Early Stage Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TH-040; NCI-2011-03308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#11-052; TH-040 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (NA-NOSE breath test) (Experimental): Patients undergo breath sample collection for the NA-NOSE breath test at baseline (2 pre-treatment samples), and post-treatment samples at regularly scheduled follow up visits, for 2 years in the absence of disease progression.
  Interventions: Procedure: breath test; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: breath test — Undergo NA-NOSE breath test
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies nanoscale artificial nose (NA-NOSE) in monitoring response and detecting recurrence after surgery or radiation therapy in patients with stage I or stage II non-small cell lung cancer (NSCLC). Using the NA-NOSE breath test may be an effective way to monitor response and detect recurrence of NSCLC after surgery or radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if a suitable fraction of patients become NA-NOSE negative within three years post treatment. We will test the hypothesis that this fraction is at most 30% versus the alternative that it is at least 50%.

SECONDARY OBJECTIVES:

I. Determine if patients who become NA-NOSE negative post treatment then become NA-NOSE positive prior to clinical recurrence.

II. Estimate the time post treatment needed to become NA-NOSE negative. III. Estimate the lead time gained between a negative to positive NA-NOSE transition and clinical recurrence.

OUTLINE:

Patients undergo breath sample collection for the NA-NOSE breath test at baseline (2 pre-treatment samples), and post treatment samples at regularly scheduled follow up visits, for 2 years in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must either have histologic or pathologically confirmed non-small cell lung cancer (NSCLC) or suspicious nodules/lesions which are going to be surgically resected before they are pathologically confirmed
* Patients must have stage I or II disease based on the parameters for staging NSCLC found in the American Joint Committee on Cancer (AJCC) cancer staging handbook seventh edition
* Patients must be deemed to be eligible candidates for either surgery or stereotactic radiation
* Stereotactic radiation treatment of stage I disease or adjuvant chemotherapy is allowed at the discretion of treating physician for the participating subject
* Patients who will have surgical resections must consent to the use of post-surgery tumor samples for correlative molecular studies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Ability to travel to appointments and willingness to participate in this study
* Ability to understand and willingness to sign a consent and Health Insurance Portability and Accountability Act (HIPAA) authorization form

Exclusion Criteria:

* Patients who have had a prior lung cancer within the last five years from the current diagnosis
* Patients having a prior malignancy within the past 3 years other than resected of basal or squamous cell carcinoma of the skin, any in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients with any prior systemic therapy for the current diagnosis of lung cancer
* Patients with a diagnosis of advanced stage disease (stage III or IV)
* Patients who are unable to comply with study and/or follow up procedures
* Patients who have uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08-23 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Successful evaluation of gas samples taken from lung cancer patients | Up to 3 years
Percent of patients that become nanoscale artificial nose negative within 3 years post-surgery | Up to 3 years
  We will test the null hypothesis that at most 30% of patients will become nanoscale artificial nose negative within 3 years post- surgery. The alternative will be that this fraction will be at least 50%. If at least 15/35 patients become nanoscale artificial nose negative within 3 years post treatment follow up we will reject the null. The test has 84.5% power and 7.31% type I error.

SECONDARY OUTCOMES:
Percentage of patients who become nanoscale artificial nose negative within 3 years and recur within that time frame that will become nanoscale artificial nose positive before recurrence | Up to 3 years
  We will test the hypothesis that at most 25% of patients who become nanoscale artificial nose negative within 3 years and recur within that time frame will become nanoscale artificial nose positive before recurrence. The alternative is that at least 50% of such patients will become nanoscale artificial nose positive before recurrence.
Time to become nanoscale artificial nose negative post treatment | Up to 3 years
  This will be done using the method of Kaplan and Meier.
Lead time between the transition from nanoscale artificial nose negativity to positivity and clinical recurrence | Up to 3 years
  We will restrict this estimate to data from patients who experience a transition and will use the method of Kaplan and Meier. We will tabulate frequencies of patients who recur with or without such a transition as well as those for patients who never become nanoscale artificial nose negative.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Borghaei, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States